CLINICAL TRIAL: NCT03312075
Title: Epidemiology and Clinical Characteristics of Non-Tuberculous Mycobacteria Infections in Cystic Fibrosis Patients.
Acronym: CIMENT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: CIMENT (29BRC17.0001)
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cystic fibrosis patients: Sputum and blood samples
  Interventions: Other: Sputum and blood samples

INTERVENTIONS:
Other: Sputum and blood samples — The cystic fibrosis patient will have a first series of sputum as well as a blood sample. On the same day of consultation, a second expectoration will be performed as far as possible.

SUMMARY:
An increase in the prevalence of infections due to non-tuberculous mycobacteria (NTM) is observed in many countries and recent data suggest the circulation of dominant clones with a possibility of human-to-human contamination. The hypothesis is made that these infections are also increasing in France and that dominant NTM clones are circulating. The last French study carried out in 2004 already showed prevalences of up to 10% in certain French regions. It is essential to know the prevalence 8 years later, taking advantage of the new recommendations for the management of patients and samples, which will homogenize practices on French territory.

No data are currently available in France on the prevalence of positive serological responses in cystic fibrosis patients. Serological analyzes of the sera collected during this study will enable us to evaluate the performance of serology in mycobacterial culture and to identify patients with no positive respiratory specimen in culture but with positive serology indicating potential contact with a mycobacterium. The establishment of a serological follow-up of these patients will allow to correlate this result with a clinical evolution and / or the detection of NTM in subsequent samples. Serology is an innovative aspect of the CIMENT study.

DETAILED DESCRIPTION:
Non-tuberculous mycobacteria (NTM) are important new pathogens in cystic fibrosis, with prevalence estimates ranging from 6% to 13%. The diagnosis of the disease in cystic fibrosis patients is difficult because the infection may remain indolent in some cases without evidence of clinical consequence, while in other patients NTM are associated with significant morbidity and mortality. Treatment requires antibiotic therapy over a prolonged period (at least 12 to 18 months) with several drugs and varies according to NTM and their antibiotic resistance profile. The development of a specialized approach (clinicians / biologists) in the management of this infection, combined with the diagnosis and treatment of NTM infections, in cystic fibrosis patients is a research priority. It is an indispensable long-term strategy for this high-risk population.

Two main elements confirm the interest of a prevalence survey of NTM infections in cystic fibrosis (CF) patients: the diagnostic difficulty of "true" infections (as opposed to simple colonizations) to NTM, and the clinical impact on respiratory functions of NTM present in these patients. Two recent contradictory studies on the impact of NTM infections in CF patients have recently been published. The German monocentric study suggests a greater deterioration of respiratory function in CF patients not infected with NTM compared to CF patients infected with NTM. 26 patients were infected with NTM: 14/26 with M. avium complex (MAC), 10/26 with M. abscessus complex and 2/26 with M. gordonae. Only 5 patients out of a dozen positive to M. abscessus and 1 in 14 positive to MAC were treated. Comparatively, the other study found a significant deterioration in respiratory function (maximum expired volume in 1 seconde) of CF patients infected with M. abscessus. This Scandinavian national study reinforced its argument by the fact that an effective treatment made it possible to find changes in maximum expired volume in 1 seconde close to that observed before the infection. Some differences are observed in these two studies; including the age of the subjects included, older in the German study, and the number of positive lung samples per patient. The German study retained the criteria of the American Thoracic Society (ATS) / Infectious Disease Society of America (IDSA) for interpreting respiratory specimens positive for MNT. However, these criteria remain very difficult to apply for CF patients because the clinical and radiological manifestations of cystic fibrosis and mycobacterial infection are confounded and other criteria are necessary, such as the number of positive pulmonary samples: 5 vs. 2 to 4 or the decline in maximum expired volume in 1 seconde in the year prior to colonization / MNT infection (-5.8% per year vs. 0.7% per year). We see here the necessity of complementary studies, in order to be able to identify the diagnostic difficulties and the impacts of the therapeutics administered in these patients. Indeed, on the one hand the therapeutic impact is very difficult to evaluate in the face of the very weak correlation between the results of the "antibiograms" and therefore in vitro and the therapeutic effect in vivo. On the other hand, precise diagnostic interpretation remains essential, as published observational studies show real discrepancies, largely due to diagnostic biases. Recently, under the auspices of the American Foundation and the European Cystic Fibrosis Society, guidelines for the management of NTM infections in CF patients have been published. To this is added the references of Microbiology.

Several authors have shown that this diagnosis is an alternative in the context of NTM infections in cystic fibrosis patients. Indeed, as mentioned above, the microbiological diagnosis is often faulted, due to the difficulty of culturing the samples and their low yield in the context of NTM infections. An indirect diagnostic approach can only reinforce the screening of cystic fibrosis patients who have had contact with a NTM. Any serological response, although unable to date an infection, is the result of a potentially protective response of the host undergoing infection, and evidence of antibodies directed against the agent's bacterial products pathogen in circulating blood. A simple colonization does not allow the appearance of antibodies. An infectious process, even inapparent, must have taken place.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of cystic fibrosis regardless of CFTR genotype
* Affiliation to the social security system
* Patients able to expectorate spontaneously
* Patients enrolled in the French Register of Cystic Fibrosis
* Minor or major patients of expectorant age
* Consent signed by the patient or the holder of parental authority for the children

Exclusion Criteria:

* Patient not registered in the French Register of Cystic Fibrosis
* Pulmonary transplant patients
* Persons deprived of liberty, persons under guardianship or curatorship, persons in emergency situations
* Person not affiliated to a social security system or not entitled

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cystic fibrosis patients
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients screened positive for NTM by the culture | 2 years
  The number of patients screened positive for NTM by the culture with regard of the number of expectorants collected will be evaluated.

SECONDARY OUTCOMES:
Number of patients screened positive for NTM by serology | 2 years
  The number of patients screened positive for NTM by serology with regard of the number of expectorants collected will be evaluated.

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - CHU Amiens, Amiens
  - CHRU Brest, Brest
  - CHU Côte de Nacre, Caen
  - CHIC Créteil, Créteil
  - CHU Grenoble, Grenoble
  - CHU Lille, Lille
  - AP-HP Hôpital Cochin, Paris
  - CHU Bordeaux, Pessac
  - Centre de Perharidy, Roscoff
  - CHU Rouen, Rouen
  - CHR Sud Réunion, Saint-Pierre
  - AP-HP Hôpital Foch, Suresnes
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours

REFERENCES:
- [Background] Qvist T, Gilljam M, Jonsson B, Taylor-Robinson D, Jensen-Fangel S, Wang M, Svahn A, Kotz K, Hansson L, Hollsing A, Hansen CR, Finstad PL, Pressler T, Hoiby N, Katzenstein TL; Scandinavian Cystic Fibrosis Study Consortium (SCFSC). Epidemiology of nontuberculous mycobacteria among patients with cystic fibrosis in Scandinavia. J Cyst Fibros. 2015 Jan;14(1):46-52. doi: 10.1016/j.jcf.2014.08.002. Epub 2014 Aug 30. PMID 25178871
- [Background] Albrecht C, Ringshausen F, Ott S, Wagner D, Rademacher J, Schneider M, Welte T, Pletz MW. Should all adult cystic fibrosis patients with repeated nontuberculous mycobacteria cultures receive specific treatment? A 10-year case-control study. Eur Respir J. 2016 May;47(5):1575-7. doi: 10.1183/13993003.01239-2015. Epub 2016 Feb 4. No abstract available. PMID 26846823
- [Background] Griffith DE, Aksamit T, Brown-Elliott BA, Catanzaro A, Daley C, Gordin F, Holland SM, Horsburgh R, Huitt G, Iademarco MF, Iseman M, Olivier K, Ruoss S, von Reyn CF, Wallace RJ Jr, Winthrop K; ATS Mycobacterial Diseases Subcommittee; American Thoracic Society; Infectious Disease Society of America. An official ATS/IDSA statement: diagnosis, treatment, and prevention of nontuberculous mycobacterial diseases. Am J Respir Crit Care Med. 2007 Feb 15;175(4):367-416. doi: 10.1164/rccm.200604-571ST. No abstract available. PMID 17277290
- [Background] Martiniano SL, Sontag MK, Daley CL, Nick JA, Sagel SD. Clinical significance of a first positive nontuberculous mycobacteria culture in cystic fibrosis. Ann Am Thorac Soc. 2014 Jan;11(1):36-44. doi: 10.1513/AnnalsATS.201309-310OC. PMID 24251858
- [Background] Floto RA, Olivier KN, Saiman L, Daley CL, Herrmann JL, Nick JA, Noone PG, Bilton D, Corris P, Gibson RL, Hempstead SE, Koetz K, Sabadosa KA, Sermet-Gaudelus I, Smyth AR, van Ingen J, Wallace RJ, Winthrop KL, Marshall BC, Haworth CS. US Cystic Fibrosis Foundation and European Cystic Fibrosis Society consensus recommendations for the management of non-tuberculous mycobacteria in individuals with cystic fibrosis: executive summary. Thorax. 2016 Jan;71(1):88-90. doi: 10.1136/thoraxjnl-2015-207983. PMID 26678435
- [Background] Jeong BH, Kim SY, Jeon K, Lee SY, Shin SJ, Koh WJ. Serodiagnosis of Mycobacterium avium complex and Mycobacterium abscessus complex pulmonary disease by use of IgA antibodies to glycopeptidolipid core antigen. J Clin Microbiol. 2013 Aug;51(8):2747-9. doi: 10.1128/JCM.00702-13. Epub 2013 Jun 5. PMID 23740728
- [Background] Qvist T, Taylor-Robinson D, Waldmann E, Olesen HV, Hansen CR, Mathiesen IH, Hoiby N, Katzenstein TL, Smyth RL, Diggle PJ, Pressler T. Comparing the harmful effects of nontuberculous mycobacteria and Gram negative bacteria on lung function in patients with cystic fibrosis. J Cyst Fibros. 2016 May;15(3):380-5. doi: 10.1016/j.jcf.2015.09.007. Epub 2015 Oct 9. PMID 26482717
- [Background] Qvist T, Pressler T, Taylor-Robinson D, Katzenstein TL, Hoiby N. Serodiagnosis of Mycobacterium abscessus complex infection in cystic fibrosis. Eur Respir J. 2015 Sep;46(3):707-16. doi: 10.1183/09031936.00011815. Epub 2015 Apr 30. PMID 25929948